CLINICAL TRIAL: NCT01892384
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BI 409306 Film-coated Tablets Given Orally q.d. for 14 Days in Patients With Schizophrenia (Randomized, Parallel-group, Double-blind, Placebo-controlled Study)
Brief Title: Safety and Tolerability of BI 409306 in Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1289.18
Record Dates: First submitted 2013-07-01; First posted 2013-07-04 (Estimated); Results first posted 2024-03-08 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — BI 409306

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BI 409306 dose 1 (Experimental): low dose, once daily
  Interventions: Drug: BI 409306
- BI 409306 dose 2 (Experimental): medium dose, once daily
  Interventions: Drug: BI 409306
- BI 409306 dose 3 (Experimental): high dose, once daily
  Interventions: Drug: BI 409306
- Placebo (Placebo Comparator): placebo, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — matching placebo
  Arms: Placebo
Drug: BI 409306 — BI 409306
  Arms: BI 409306 dose 1; BI 409306 dose 2; BI 409306 dose 3

SUMMARY:
The primary objective of the current study is to investigate the safety and tolerability of BI 409306 in schizophrenic patients following oral administration of multiple low, medium, and high doses over 14 days.

A secondary objective is the exploration of the pharmacokinetics and pharmacodynamics of BI 409306 in schizophrenic patients.

ELIGIBILITY:
Inclusion criteria:

1. Patients with established diagnoses of schizophrenia (per Diagnostic and Statistical Manual of Mental Disorders (DSM-IV)) with the following clinical features:

   1. Clinically stable and are in the residual (non-acute) phase of their illness for at least 8 weeks.
   2. Maintained on current antipsychotic medications and current dose for at least 8 weeks.
   3. Have no more than a moderate severity rating on hallucinations and delusions (e.g. Brief Psychiatric Rating Scale (BPRS) Hallucinatory Behavior or Unusual Thought Content item score < or =4).
   4. Have no more than a moderate severity rating on positive formal thought disorder (e.g. BPRS Conceptual Disorganization item score < or =4).
   5. Have no more than a moderate severity rating on negative symptoms (Positive and Negative Syndrome Scale negative syndrome total score <15).
   6. Have a minimal level of extrapyramidal symptoms (e.g. Simpson-Angus Scale total score < 6) and depressive symptoms (e.g. Calgary Depression Scale total score < 10).
2. Male or female patients age > or = 18 and < or =55 years.
3. Patients must exhibit reliability and physiologic capability to comply with all protocol procedures.
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation. If the patient needs a legal representative, then this legal representative must give written consent as well.

Exclusion criteria:

1. Patient treated with more than one antipsychotic or not stabilized on antipsychotic treatment, or having had electroconvulsive therapy within the last 30 days
2. Patient's cognitive impairment severity compromises the validity of the cognitive outcome measures, in the clinical judgment of the investigator.
3. Any suicidal behavior in the past 2 years (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior).
4. Any suicidal ideation of type 4 or 5 in the Columbia Suicidal Severity Rating Scale (C-SSRS) in the past 3 months (i.e. active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent).
5. Any finding of the medical examination (including BP, PR and ECG) or laboratory value deviating from normal and of clinical relevance in the judgment of the investigator.
6. Any evidence of a clinically relevant concomitant disease.
7. History or diagnosis of symptomatic and unstable/uncontrolled gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, haematological or hormonal disorders.
8. Female patients that are of child-bearing potential or currently breastfeeding.
9. Known history, or new diagnosis per screening labs, of HIV infection.
10. History of neurologic (e.g. stroke, seizure without a clear and resolved etiology, concussion accompanying loss of consciousness) or psychiatric condition that the investigator deems may interfere with interpretability of data
11. History of malignancy within the last 5 years, except for basal cell carcinoma.
12. Planned elective surgery requiring general anaesthesia, or hospitalisation for more than 1 day during the study period.
13. Any other clinical condition that, in the opinion of the investigator, would jeopardize a patient's safety while participating in this clinical trial.
14. Significant history of drug dependence or abuse (including alcohol, as defined in Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) or in the opinion of the investigator) within the last two years prior to informed consent, or a positive urine drug screen for cocaine, opioid, phencyclidine (PCP), amphetamine or marijuana at screening.
15. Participation in another trial with an investigational drug or procedure within 30 days prior to screening or previous participation in any BI 409306 study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-06-28 (Actual); Primary Completion 2013-12-05 (Actual); Study Completion 2013-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1289.18.1 Boehringer Ingelheim Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Brown D, Daniels K, Pichereau S, Sand M. A Phase IC Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Cognitive Outcomes of BI 409306 in Patients with Mild-to-Moderate Schizophrenia. Neurol Ther. 2018 Jun;7(1):129-139. doi: 10.1007/s40120-017-0085-5. Epub 2017 Nov 24. PMID 29177699
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, double-blind, parallel-group, placebo-controlled trial in patients with mild-to-moderate schizophrenia. Patients were enrolled in the study once informed consent had been obtained. Patients who subsequently met all eligibility criteria at screening were randomized in a 1:1:1:1 ratio to one of four treatment groups.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 409306 25mg: Patients received BI 409306 25mg (low dose), administered orally, once daily for 14 days
- BI 409306 50mg: Patients received BI 409306 50mg (medium dose), administered orally, once daily for 14 days
- BI 409306 100mg: Patients received BI 409306 100mg (high dose), administered orally, once daily for 14 days
- Placebo: Patients received placebo, administered orally, once daily for 14 days
Period: Overall Study
Arm/Group | BI 409306 25mg | BI 409306 50mg | BI 409306 100mg | Placebo
Started | 10 | 10 | 10 | 10
Completed | 9 | 9 | 10 | 10
Not Completed | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set which included all randomized patients who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 409306 25mg | BI 409306 50mg | BI 409306 100mg | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.9 (9.5) | 42.5 (9.0) | 42.5 (8.4) | 37.8 (9.5) | 40.2 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 0 | 2 | 5
  Male | 10 | 7 | 10 | 8 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 2 | 2 | 9
  Not Hispanic or Latino | 9 | 6 | 8 | 8 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 7 | 5 | 21
  White | 5 | 6 | 3 | 5 | 19
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Drug-related Adverse Events
Description: Number of participants with drug-related adverse events.
Time Frame: From first drug administration until 30 days after last drug administration, up to 44 days.
Population: Treated set which included all randomized patients who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | BI 409306 25mg | BI 409306 50mg | BI 409306 100mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
Participants | 1 | 3 | 2 | 3

2. Secondary Outcome: Maximum Measured Concentration of BI 409306 in Plasma After Single Dose (Cmax)
Description: Maximum measured concentration of BI 409306 in plasma after single dose (Cmax) is presented.
Time Frame: 2 hours (h) before first drug administration and 10minutes (min), 20min, 30min, 45min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h and 14h after first drug administration
Population: Pharmacokinetic (PK) set which included all participants who received at least one dose of BI 409306 and had no important protocol violations relevant to the evaluation of PK and provided at least one evaluable observation for a PK endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Litre (nmol/L)
Arm/Group | BI 409306 25mg | BI 409306 50mg | BI 409306 100mg
Number analyzed (Participants) | 10 | 10 | 10
nanomole/Litre (nmol/L) | 138 (91.9) | 431 (73.3) | 998 (106.0)

3. Secondary Outcome: Maximum Measured Concentration of BI 409306 in Plasma at Steady-state (Cmax,ss)
Description: Maximum measured concentration of BI 409306 in plasma at steady-state (Cmax,ss) is presented.
Time Frame: 2 hours (h) before drug administration and 10minutes (min), 20min, 30min, 45min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 14h, 24h, 48h and 72h after drug administration on day 14.
Population: Pharmacokinetic (PK) set which included all participants who received at least one dose of BI 409306 and had no important protocol violations relevant to the evaluation of PK and provided at least one evaluable observation for a PK endpoint. Two patients were discontinued from treatment after 6 days (25 mg group) or 5 days (50 mg group) after withdrawing consent.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Litre (nmol/L)
Arm/Group | BI 409306 25mg | BI 409306 50mg | BI 409306 100mg
Number analyzed (Participants) | 9 | 9 | 10
nanomole/Litre (nmol/L) | 99.2 (86.8) | 631 (90.9) | 1290 (74.4)

4. Secondary Outcome: Time From Dosing to Maximum Measured Concentration of BI 409306 in Plasma After Single Dose (Tmax)
Description: Time from dosing to maximum measured concentration of BI 409306 in plasma after single dose (tmax) is presented.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | BI 409306 25mg | BI 409306 50mg | BI 409306 100mg
Number analyzed (Participants) | 10 | 10 | 10
Hours | 0.625 [0.33 to 1.50] | 0.625 [0.33 to 2.00] | 0.750 [0.33 to 2.00]

5. Secondary Outcome: Time From Dosing to Maximum Measured Concentration of BI 409306 in Plasma at Steady-state (Tmax,ss)
Description: Time from dosing to maximum measured concentration of BI 409306 in plasma at steady-state (tmax,ss) is presented.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | BI 409306 25mg | BI 409306 50mg | BI 409306 100mg
Number analyzed (Participants) | 9 | 9 | 10
Hours | 0.750 [0.33 to 1.00] | 0.333 [0.33 to 1.50] | 0.625 [0.33 to 1.50]

6. Secondary Outcome: Area Under the Concentration-time Curve of BI 409306 in Plasma Over the Time Interval From 0 Extrapolated to Infinity After a Single Dose (AUC0-infinity)
Description: Area under the concentration-time curve of BI 409306 in plasma over the time interval from 0 extrapolated to infinity after a single dose (AUC0-infinity) is presented.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole*hour/Litre (nmol*h/L)
Arm/Group | BI 409306 25mg | BI 409306 50mg | BI 409306 100mg
Number analyzed (Participants) | 10 | 10 | 10
nanomole*hour/Litre (nmol*h/L) | 217 (107.0) | 770 (98.4) | 2020 (108.0)

7. Secondary Outcome: Area Under the Concentration-time Curve of BI 409306 in Plasma at Steady State Over a Uniform Dosing Interval Tau (AUCtau,ss)
Description: Area under the concentration-time curve of BI 409306 in plasma at steady state over a uniform dosing interval tau (AUCtau,ss) is presented.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole*hour/Litre (nmol*h/L)
Arm/Group | BI 409306 25mg | BI 409306 50mg | BI 409306 100mg
Number analyzed (Participants) | 9 | 9 | 10
nanomole*hour/Litre (nmol*h/L) | 147 (112.0) | 969 (104.0) | 2280 (86.8)

ADVERSE EVENTS:
Time Frame: From first dose of study medication until 30 days after the last dose of study medication, up to 44 days.
Description: Treated set which included all randomized patients who received at least one dose of study medication.
Groups:
- Total.: All patients entered into the study received either BI 409306 or placebo once daily for 14 days.
Arm/Group | BI 409306 25mg | BI 409306 50mg | BI 409306 100mg | Placebo | Total.
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/40
Other Adverse Events (participants affected / at risk) | 4/10 | 9/10 | 6/10 | 4/10 | 23/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 409306 25mg (N=10) | BI 409306 50mg (N=10) | BI 409306 100mg (N=10) | Placebo (N=10) | Total. (N=40)
Photopsia (Eye disorders) | 0 | 1 | 1 | 0 | 2
Vision blurred (Eye disorders) | 2 | 3 | 1 | 2 | 8
Visual impairment (Eye disorders) | 1 | 1 | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 0 | 1
Pre-existing condition improved (General disorders) | 0 | 0 | 0 | 1 | 1
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 2
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Visual field defect (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.